CLINICAL TRIAL: NCT00002107
Title: A Phase I Study of Subcutaneously Administered Proleukin (Aldesleukin) in HIV-Infected Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chiron Corporation (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 085A; CS-L293-09
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1995-03

CONDITIONS: HIV Infections
Keywords: Interleukin-2; Acquired Immunodeficiency Syndrome; AIDS-Related Complex
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — aldesleukin

INTERVENTIONS:
Drug: Aldesleukin

SUMMARY:
To determine the MTD and dose-limiting toxicities of recombinant interleukin-2 (aldesleukin; Proleukin) administered subcutaneously in HIV-seropositive patients. To identify a tolerable subcutaneous regimen that will replicate the immunologic improvement demonstrated in the outpatient polyethylene glycolated IL-2 and high-dose continuous infusion IL-2 studies. To evaluate the incidence and level of anti-IL-2 antibody formation to subcutaneously administered Proleukin in this patient population.

DETAILED DESCRIPTION:
Patients will receive subcutaneous Proleukin, and the MTD will be determined.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Documented HIV infection by ELISA and Western blot.
* CD4 count > 200 cells/mm3.

Required:

* FDA-approved antiretroviral therapy for at least 2 months prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Davies Med Ctr / c/o HIV Institute, San Francisco, California, United States

REFERENCES:
- [Background] Follansbee SE, Lacarrubba S, Fyfe G. Dose-ranging study of interleukin II (IL-2) in HIV-infected men on antiretroviral therapy (ARV). Conf Retroviruses Opportunistic Infect. 1997 Jan 22-26;4th:142 (abstract no 419)